CLINICAL TRIAL: NCT00771472
Title: Phase I Clinical Study of MK-0683 in Patients With Relapsed or Refractory Cutaneous T-Cell Lymphoma (CTCL)
Brief Title: Vorinostat (MK-0683) Phase I Study in Cutaneous T-Cell Lymphoma (CTCL) Patients (MK-0683-089 EXT1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0683-089; 2008_565
Record Dates: First submitted 2008-10-09; First posted 2008-10-13 (Estimated); Results first posted 2012-07-04 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vorinostat (Experimental)
  Interventions: Drug: vorinostat

INTERVENTIONS:
Drug: vorinostat — Parts I & II: Vorinostat (400 mg) Oral, daily (QD). Treatment period is 28 days per cycle.
  Other Names: MK-0683; Zolinza

SUMMARY:
Part I evaluates the safety, tolerability and pharmacokinetics (PK) of vorinostat in Japanese patients with relapsed or refractory CTCL. Part II evaluates the safety of vorinostat in Japanese pts. with relapsed or refractory CTCL. Relapsed or refractory CTCL patients will be newly enrolled in Part II.

ELIGIBILITY:
Inclusion Criteria (Parts I & II):

* Patients With CTCL Who Have Progressive, Persistent Or Recurrent Disease Subsequent To At Least One Prior Therapy
* Eastern Cooperative Oncology Group (ECOG) Performance Status Must Be 0-2
* Patients Have Adequate Bone Marrow, Liver Function And Renal Function

Exclusion Criteria (Parts I & II):

* Patients Had Prior Therapy Within 3 Weeks Before Registration, Or Have Not Recovered From Toxicities Of Prior Therapy
* Patients Have Uncontrolled Intercurrent Illness
* Pregnant Or Women Have A Will To Be Pregnant And Lactating Woman

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Wada H, Tsuboi R, Kato Y, Sugaya M, Tobinai K, Hamada T, Shimamoto T, Noguchi K, Iwatsuki K. Phase I and pharmacokinetic study of the oral histone deacetylase inhibitor vorinostat in Japanese patients with relapsed or refractory cutaneous T-cell lymphoma. J Dermatol. 2012 Oct;39(10):823-8. doi: 10.1111/j.1346-8138.2012.01554.x. Epub 2012 Apr 16. PMID 22506596

RESULTS

PARTICIPANT FLOW:
Groups:
- Part I; Part II: Vorinostat 400 mg oral, daily (QD). Treatment period was 28 days per cycle.
Period: Overall Study
Arm/Group | Part I | Part II
Started | 6 | 4
Completed | 0 | 0
Not Completed | 6 | 4
Not completed — Physician Decision | 2 | 3
Not completed — Progressive Disease | 3 | 1
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Vorinostat: Parts I & II: vorinostat (400 mg) oral, daily (QD). Treatment period was 28 days per cycle.
Arm/Group | Vorinostat
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Region of Enrollment [Number; unit: participants]
  Japan | 10

OUTCOME MEASURES:

1. Primary Outcome: Parts I & II: Number of Participants Experiencing Clinical or Laboratory Adverse Experiences (AE)
Description: A laboratory AE is defined as any unfavorable & unintended change in the chemistry of the body temporally associated with the use of study product, whether or not considered related to the use of the product. A clinical AE is defined similarly but also includes changes in structure or function of the body.
Time Frame: Day 1 up until 30 days post study completion or early termination (up to approximately 506 days)
Measure: Number; unit: participants
Arm/Group | Vorinostat
Number analyzed (Participants) | 10
participants
  Clinical AEs | 10
  Laboratory AEs | 6

2. Secondary Outcome: Part I: Total Drug Exposure (Area Under the Concentration Curve, AUC[0-24 Hours])
Description: Blood samples taken as follows:
  Day 1 & Day 28 of Cycle 1: pre dose, and 0.25, 0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 10, 12 and 24 hours after dosing of vorinostat.
Time Frame: Days 1 & 28 of Cycle 1
Population: Number of participants with samples at the specified time point
Measure: Geometric Mean (Standard Deviation); unit: µM*hr
Groups:
- Vorinostat: Part I: vorinostat (400 mg) oral, daily (QD). Treatment period was 28 days per cycle.
Arm/Group | Vorinostat
Number analyzed (Participants) | 6
µM*hr
  Day 1 (n=6) | 4.59 (2.34)
  Day 28 (n=5) | 5.59 (1.24)

3. Primary Outcome: Part I: Number of Participants Experiencing Dose Limiting Toxicity (DLT)
Description: A DLT was defined as any of the following (per Common Terminology Criteria for Adverse Events [CTCAE] version 3.0):
  * Grade 3 (severe)-4 (life-threatening) neutropenia with fever ≥ 38.5ºC
  * Grade 3-4 neutropenia with an infection requiring antibiotic or antifungal treatment
  * Grade 4 neutropenia lasting at least 5 days
  * Grade 4 thrombocytopenia
  * Other Grade 4 hematologic toxicity, including a decrease in hemoglobin, only at the discretion of the principal investigator
  * Grade 3 or 4 non-hematologic event, except which are manageable by supportive care or non-prohibited therapies
Time Frame: Day 1 to Day 28
Measure: Number; unit: participants
Arm/Group | Vorinostat
Number analyzed (Participants) | 6
participants | 1

4. Secondary Outcome: Part I: Maximum Drug Concentration (Cmax)
Description: as for outcome 2
Time Frame: Days 1 & 28 of Cycle 1
Population: Number of participants with samples at the specified time point
Measure: Geometric Mean (Standard Deviation); unit: µM
Arm/Group | Vorinostat
Number analyzed (Participants) | 6
µM
  Day 1 (n=6) | 0.83 (0.37)
  Day 28 (n=5) | 1.17 (0.37)

5. Secondary Outcome: Part I: Time at Which Cmax Occurs (Tmax)
Description: as for outcome 2
Time Frame: Days 1 & 28 of Cycle 1
Population: Number of participants with samples at the specified time point
Measure: Median (Full Range); unit: hours
Arm/Group | Vorinostat
Number analyzed (Participants) | 6
hours
  Day 1 (n=6) | 2.91 [2.00 to 6.00]
  Day 28 (n=5) | 3.73 [2.93 to 4.28]

6. Secondary Outcome: Part I: The Amount of Time it Takes for the Drug Concentration to Decrease by Half (T1/2)
Description: as for outcome 2
Time Frame: Days 1 & 28 of Cycle 1
Population: Number of participants with samples at the specified time point
Measure: Geometric Mean (Standard Deviation); unit: hours
Arm/Group | Vorinostat
Number analyzed (Participants) | 6
hours
  Day 1 (n=5) | 1.94 (1.30)
  Day 28 (n=4) | 2.30 (1.10)

ADVERSE EVENTS:
Groups:
- Vorinostat: Parts I & II: vorinostat(400 mg) Oral, daily (QD). Treatment period was 28 days per cycle.
Arm/Group | Vorinostat
Serious Adverse Events (participants affected / at risk) | 3/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat (N=10)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Cellulitis streptococcal (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat (N=10)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
Erythropenia (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 3 (7)
Lymphopenia (Blood and lymphatic system disorders) | 2 (3)
Neutropenia (Blood and lymphatic system disorders) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (29)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Vitreous floaters (Eye disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (3)
Cheilitis (Gastrointestinal disorders) | 2 (4)
Constipation (Gastrointestinal disorders) | 3 (6)
Diarrhoea (Gastrointestinal disorders) | 4 (5)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (16)
Vomiting (Gastrointestinal disorders) | 4 (7)
Chills (General disorders) | 1 (2)
Fatigue (General disorders) | 4 (6)
Malaise (General disorders) | 5 (10)
Oedema peripheral (General disorders) | 2 (2)
Pyrexia (General disorders) | 4 (9)
Swelling (General disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (3)
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 (14)
Bacterial infection (Infections and infestations) | 1 (1)
Body tinea (Infections and infestations) | 1 (1)
Candidiasis (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Keratitis herpetic (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (3)
Aspartate aminotransferase increased (Investigations) | 2 (5)
Blood alkaline phosphatase increased (Investigations) | 1 (2)
Blood cholinesterase increased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 2 (3)
Blood fibrinogen increased (Investigations) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (3)
Blood urea increased (Investigations) | 1 (1)
C-reactive protein increased (Investigations) | 1 (2)
Fibrin D dimer increased (Investigations) | 1 (2)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (2)
Prothrombin time shortened (Investigations) | 1 (1)
Weight decreased (Investigations) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 6 (11)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Hypercreatininaemia (Metabolism and nutrition disorders) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (7)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesaemia (Metabolism and nutrition disorders) | 4 (6)
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 (3)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 4 (7)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 2 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Ageusia (Nervous system disorders) | 1 (1)
Dizziness postural (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 4 (5)
Headache (Nervous system disorders) | 3 (5)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 2 (2)
Somnolence (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Haemoglobinuria (Renal and urinary disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 4 (4)
Renal impairment (Renal and urinary disorders) | 2 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (12)
Hypotension (Vascular disorders) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication guidelines.